CLINICAL TRIAL: NCT00794183
Title: A Pilot Study of theRelationship Between Atrio-Ventricular Delay and Changes in Biochemical Markers of Chronic Heart Failure During Cardiac Resynchronization Therapy (BRAVO-CRT)
Brief Title: A Pilot Study Comparing the Programmed Delay Between the Atrial and Ventricle Interval
Acronym: BRAVO-CRT
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: funding difficulty
Sponsor: University of Minnesota (Other)
Collaborators: Minnesota Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0303M44604
Record Dates: First submitted 2008-11-18; First posted 2008-11-19 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Heart Failure
Keywords: heart failure; CRT; CHF
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): AVD set by taking the larger of 0.50ms or A-V interval 0.30
  Interventions: Device: CRT device settings
- 2 (Active Comparator): AVD set by taking the larger of 0.50ms or A-V interval 0.50
  Interventions: Device: CRT device settings
- 3 (Active Comparator): AVD set by taking the larger of 0.50ms or A-V interval 0.70
  Interventions: Device: CRT device settings

INTERVENTIONS:
Device: CRT device settings — Comparision of A-V delay settings

SUMMARY:
The idea of this study is to compare different ways of setting up a pacemaker, using blood tests to give us information about how well it's working. We hope to learn if we can use this approach to figure out the best pacemaker setup ("programming") for each individual patient.

The setting we propose to adjust is the timing between the impulse sent between top and bottom chambers.

DETAILED DESCRIPTION:
There are different kinds of pacemakers and different ways they can be set up to try to make the heart beat regularly. A normal heart has four chambers; these four chambers pump in a co-ordinated way to move blood effectively. When pacemakers were first invented, they told the heart when to pump, but didn't make the four chambers work well together. Newer pacemakers can give more detailed instructions, so the chambers work together more effectively. We already know that the newer (bi-ventricular) pacemakers work better for some patients with heart failure.

There are blood tests (often referred to as "markers") that give us information about how well your heart is working and about how your body is responding to heart failure. The idea of this study is to compare different ways of setting up a pacemaker, using these blood tests to give us information about how well it's working. We hope to learn if we can use this approach to figure out the best pacemaker setup ("programming") for each individual patient.

Usually pacemakers have two wires or leads, one is in the top right chamber and the other in the bottom right chamber of the heart. The newer pacemakers, which are given to patients with heart failure, have an additional lead or wire, which goes to the left side of the heart. So when heart contracts the lead from top chamber sends impulses to bottom chambers and the leads in right and left sides of bottom chamber responds by sending impulses in a co-ordinated way enabling heart to contract efficiently.

Currently, the standard way of treating patients with heart failure is by pacing the top and then bottom chambers, based on a timing interval determined by ultrasound, while also pacing the two bottom chambers in a coordinated manner. There are differences of opinion among experts and by previous studies regarding this method. Pacing is accomplished through pacemaker wires, which are placed in the right top chamber, the right bottom chamber and the left bottom chamber of the heart.

The setting we propose to adjust is the timing between the impulse sent between top and bottom chambers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic heart failure
* patients on stable pharmacologic therapy for at least 3 months
* EF< 35%
* age >18 years
* NYHA functional class III or IV
* eligible for either CRT pacer or CRT defibrillator for heart failure
* Ischemic or non-ischemic cardiomyopathy
* patients that are able to tolerate VDD mode with a lower rate of 40bpm programming

Exclusion Criteria:

* systolic blood pressure <70mmHg
* Likely to receive a left ventricular assist device or cardiac transplant within 6 months of implant procedure
* patients who have previously received a CRT device
* documented atrial fibrillation
* complete heart block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2004-06; Primary Completion 2010-05 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To assess the effect of CRT atrioventricular delay settings on biochemical markers in blood through 6 months | end of the study

SECONDARY OUTCOMES:
assess effects of echocardiogram through 6months after CRT on heart failure | end to study
assess the effects of minnesota Living with heart failure questionaire through 6 months after CRT on heart failure | end of study
assess effects of six minute hall walk through 6 months after CRt on heart failure | end of study
assess effects of SDANN through 6 months after CRT on heart failure | end of study

CONTACTS AND LOCATIONS:
Overall Officials: David G Benditt, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States